CLINICAL TRIAL: NCT04105062
Title: Evaluation of LS301 Uptake in Tumors of Patients Undergoing Liver, Pancreas, or Gastric Surgery
Brief Title: LS301 Uptake in Tumors of Patients Undergoing Liver, Pancreas, or Gastric Surgery
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: One of the investigators is leaving the University.
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Diagnostic
Other Study IDs: 201911165
Record Dates: First submitted 2019-09-20; First posted 2019-09-26 (Actual); Last update posted 2021-12-09 (Actual); Status verified 2021-12

CONDITIONS: Pancreatic Cancer; Liver Cancer; Gastric Cancer; Gastrointestinal Stromal Cancer; Metastatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms; Liver Neoplasms; Stomach Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Intervention Model Description: A rolling six design will be used to enroll patients in the phase 1 dose escalating portion of the study, during which LS301 will be administered intravenously at one of three doses. After the optimal dose has been determined, an additional 9 patients will be enrolled in the phase I expansion cohort to evaluate for safety. The optimal imaging dose of LS301 determined in phase I will be administered in 88 patients in the phase II portion of the study.
Who Masked: Care Provider
Masking Description: The operating surgeon will remain blinded to the fluorescence images throughout the operation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (4):
- Phase I: LS301 Dose Level 1 (0.05 mg/kg) (Experimental): * The patient will undergo intravenous injection of LS301 4-24 hours prior to surgery.
  * The operating surgeon will conduct surgery as usual without using a device to visualize LS301 fluorescence. To prevent bias in data acquisition, a second surgeon will wear the CVG at the completion of the surgery to examine the excised tissue at the surgical margins and the surgical resection bed.
  * The operating surgeon will remain blinded to the fluorescence images throughout the operation. The examining surgeon will wear the CVG and image all six anatomical aspects (superior, inferior, anterior, posterior, medial and lateral) of the surgical specimen as well as the surgical cavity for LS301 fluorescence.
  Interventions: Drug: LS301; Device: Cancer Vision Goggles
- Phase I: LS301 Dose Level 2 (0.075 mg/kg) (Experimental): * The patient will undergo intravenous injection of LS301 4-24 hours prior to surgery.
  * The operating surgeon will conduct surgery as usual without using a device to visualize LS301 fluorescence. To prevent bias in data acquisition, a second surgeon will wear the CVG at the completion of the surgery to examine the excised tissue at the surgical margins and the surgical resection bed.
  * The operating surgeon will remain blinded to the fluorescence images throughout the operation. The examining surgeon will wear the CVG and image all six anatomical aspects (superior, inferior, anterior, posterior, medial and lateral) of the surgical specimen as well as the surgical cavity for LS301 fluorescence.
  Interventions: Drug: LS301; Device: Cancer Vision Goggles
- Phase I: LS301 Dose Level 3 (0.1 mg/kg) (Experimental): * The patient will undergo intravenous injection of LS301 4-24 hours prior to surgery.
  * The operating surgeon will conduct surgery as usual without using a device to visualize LS301 fluorescence. To prevent bias in data acquisition, a second surgeon will wear the CVG at the completion of the surgery to examine the excised tissue at the surgical margins and the surgical resection bed.
  * The operating surgeon will remain blinded to the fluorescence images throughout the operation. The examining surgeon will wear the CVG and image all six anatomical aspects (superior, inferior, anterior, posterior, medial and lateral) of the surgical specimen as well as the surgical cavity for LS301 fluorescence.
  Interventions: Drug: LS301; Device: Cancer Vision Goggles
- Phase II: LS301 Dose determined in Phase I (Experimental): * The patient will undergo intravenous injection of LS301 4-24 hours prior to surgery.
  * The operating surgeon will conduct surgery as usual without using a device to visualize LS301 fluorescence. To prevent bias in data acquisition, a second surgeon will wear the CVG at the completion of the surgery to examine the excised tissue at the surgical margins and the surgical resection bed.
  * The operating surgeon will remain blinded to the fluorescence images throughout the operation. The examining surgeon will wear the CVG and image all six anatomical aspects (superior, inferior, anterior, posterior, medial and lateral) of the surgical specimen as well as the surgical cavity for LS301 fluorescence.
  Interventions: Drug: LS301; Device: Cancer Vision Goggles

INTERVENTIONS:
Drug: LS301 — -LS301 is produced at the Optical Radiology Laboratory at Washington University School of Medicine
Device: Cancer Vision Goggles — -Non-significant risk device
  Other Names: CVG

SUMMARY:
The preclinical data have demonstrated the feasibility of fluorescence-guided tumor resection by the Cancer Vision Googles (CVG) with LS301 in animal models. In this study, the investigators will conduct intraoperative imaging procedures that have minimal interference with ongoing surgery. The underlying hypothesis is that the accurate detection of all cancer cells highlighted by LS301 during surgery will reduce the number of patients with margin positivity to less than 5%, compared to the current surgical paradigm of greater than 15% in pancreatic cancer, for example. The pilot study will obtain critical data required to address the larger question of surgical margin assessment in a full Phase I clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed patients with gastrointestinal cancers, including pancreas, liver, gastric cancer, gastrointestinal stromal tumors, and metastatic cancers undergoing surgical resection as standard of care treatment.
* At least 18 years of age.
* For the first cohort of patients enrolled, must have an ECG with no prolonged intervals.
* Able to understand and willing to sign a written informed consent document.

Exclusion Criteria:

* Contraindications for surgery.
* Receiving any investigational agents.
* History of allergic reactions attributed to ICG or other agents used in the study, include known iodide or seafood allergy. We do not expect many of these adverse reactions with LS301 because it is not radioactive and does not possess iodinated counterions.
* Presence of underlying lung disease.
* Pregnant. Female patients of childbearing potential must have a negative serum or urine pregnancy test no more than 7 days before start of participation.
* Breastfeeding. Patients who are breastfeeding are excluded from this study because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with LS301.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-12-31 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Phase I only: Safety of LS301 as measured by incidence of related adverse events per patient | From time of injection to 1 hour post-injection
  * Safety evaluation includes vital signs, clinical laboratory testing and ECG, measured pre- (within 10-15 minutes or 30 minutes of injection) and post-injection (within 30 minutes or/and at ~60 minutes).
  * Adverse events will be graded using NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5.0
Phase I only: Optimal imaging dose of LS301 | From time of injection to 1 hour post-injection
  * The optimal will be the dose at which fewer than 2 dose-limiting toxicities (DLTs) are observed and optimal image quality is observed. It need not be the maximum tolerated dose (MTD) if optimal image quality is observed at a lower dose than the MTD
  * DLT is defined as any grade 2 or above toxicity that occurs during the hour after injection that is considered possibly, probably, or definitely related to LS301.
Phase II only: Ability of LS301 to predict presence of positive margins | At the time of pathological analysis (within 2-3 days of surgery)
  * Margin status called by LS301 and CVG will be compared to the gold standard histopathological results
  * The histopathological results of margin positivity has the following possible results: margin negative, margin positive at LS301 and CVG identified locations, margin positive at LS301 and CVG unidentified locations. Using LS301 and CVG, the exercised tissue will be considered to be margin positive and have ink marked at the identified locations if any positive margins are observed; otherwise, the margin is considered negative.

CONTACTS AND LOCATIONS:
Overall Officials: Ryan C Fields, M.D., Principal Investigator — Washington University School of Medicine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu